CLINICAL TRIAL: NCT01284400
Title: The Japanese Heart Failure Outpatients Disease Management and Cardiac Evaluation (J-HOMECARE)
Brief Title: Home-based Disease Management Program to Improve Clinical Outcomes in Patients With Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japanese Heart Failure Outpatient Disease Management Evaluation Investigators (Network)
Responsible Party: Hiroyuki Tsutsui, Department of Cardiovascular Medicine, Hokkaido University Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J-HOMECARE; UMIN000000565 (Other: University hospital Medical Information Network)
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Heart Failure
Keywords: heart failure; disease management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disease management (Experimental)
  Interventions: Other: Home-based disease management
- Usual treatment and care (No Intervention)

INTERVENTIONS:
Other: Home-based disease management — Symptom monitoring, comprehensive advice, and counseling at home by nurses, as well as telephone follow-up by nurses
  Arms: Disease management

SUMMARY:
Although many studies have demonstrated the efficacy of disease management programs on mortality, morbidity, quality of life (Qol), and medical cost in patients with heart failure (HF), no study has focused on psychological status as an outcome of disease management in patients with HF. Disease management could lead to the reduction of psychological distress, thus improving the self-care ability and adherence of patients with HF. In addition, very little information is available on the effectiveness of disease management programs in areas other than the US and Europe.The Japanese Heart Failure Outpatients Disease Management and Cardiac Evaluation (J-HOMECARE) has designed a randomized controlled trial to evaluate the efficacy of home-based disease management programs compared with usual care in improving psychosocial status, mortality, HF hospitalization, and Qol in Japanese HF patients.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years

Exclusion criteria

1. End-stage HF defined as requiring mechanical support or continues intravenous inotropic support
2. A serious life-threatening illness with a life-expectancy of <6 months Within the past 3 months
3. Cognitive dysfunction
4. Substance abuse or psychotic disorder
5. Managed by visiting nursing
6. Long distance between patients' home and hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Psychosocial status (depression, anxiety) | up to 12 months

SECONDARY OUTCOMES:
Death | up to 12 months
Readmission due to heart failure | up to 12 months
Hospital admission | up to 12 months
Quality of life | up to 12 months
Physical activity | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Tsutsui, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Hokkaido University Graduate School of Medicine

REFERENCES:
- [Derived] Tsuchihashi-Makaya M, Matsuo H, Kakinoki S, Takechi S, Kinugawa S, Tsutsui H; J-HOMECARE Investigators. Home-based disease management program to improve psychological status in patients with heart failure in Japan. Circ J. 2013;77(4):926-33. doi: 10.1253/circj.cj-13-0115. Epub 2013 Mar 15. PMID 23502992
- [Derived] Tsuchihashi-Makaya M, Matsuo H, Kakinoki S, Takechi S, Tsutsui H; J-HOMECARE Investigators. Rationale and design of the Japanese heart failure outpatients disease management and cardiac evaluation (J-HOMECARE). J Cardiol. 2011 Sep;58(2):165-72. doi: 10.1016/j.jjcc.2011.04.004. PMID 21640556